CLINICAL TRIAL: NCT02848534
Title: The Value of the Neutrophil to Lymphocyte Ratio in the Diagnosis of Bacterial Infections
Acronym: RNL-MI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-40 Schmidt-2
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Bacterial Infections
Keywords: fever; hyperthermia; inflammatory syndrome
MeSH Terms: conditions — Bacterial Infections; Fever; Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Biological: neutrophil to lymphocyte ratio — value of the neutrophil to lymphocyte ratio in the diagnosis of bacterial infections

SUMMARY:
The "gold standard" for diagnosing a bacterial infection is isolation of the pathogenic germ, which is not easy in routine clinical practice.

Conventional markers do not have sufficient diagnostic value for making a rapid diagnosis on admission. A 2004 literature calculated the diagnostic values of C-reactive protein (CRP) and procalcitonin (PCT) levels for the diagnosis of bacterial infections, relative to other causes of inflammation. For CRP, the sensitivity was 75% (95% CI: 62%-84%) and the specificity was 67% (95% CI: 56%-77%). For PCT, the sensitivity was 88% (95% CI: 62%-84%) and the specificity was 81% (95% CI: 67%-90%).

The first cellular immune response to infection consists of the mobilization of polynuclear neutrophils from the bone marrow to the infection site under the effect of pre-inflammatory cytokines, as well as the apoptosis of lymphocytes and their sequestration at the infection site. This results in lymphopenia and the elevated polynuclear neutrophil count (PNN) observed in bacterial infections.

Hence, it is legitimate to hypothesize that the neutrophil to lymphocyte ratio (NLR) can be used in the diagnosis of bacterial infection. This ratio's value in the diagnosis of sepsis in the emergency department was studied and the researchers found higher diagnostic values than for CRP and PCT.

The NLR's potential value in the diagnosis of a bacterial infection in a context of fever or hyperthermia (regardless of the presence or absence of bacteraemia) has not been studied before. This ratio could also be compared with standard biomarkers (CRP and PCT levels, the white blood cell count and the PNN).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted for fever/inflammatory syndrome to the internal medicine department at Amiens University Hospital between January 1 st 2011 and December 31 st 2014 (hyperthermia > 38°5 and/or inflammatory syndrome, defined as an increase in CRP >10 mg/L).

Exclusion Criteria:

* Known conditions or treatments that may influence the blood count (haematological and neoplastic diseases, seropositivity for HIV, chemotherapy, and corticotherapy).
* Pregnancy.
* A course of antibiotics administered in the 48 hours before the
* blood count (risk of sample negativity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted for fever/inflammatory syndrome to the internal medicine department at Amiens University Hospital between January 1 st 2011 and December 31 st 2014 (hyperthermia > 38°5 and/or inflammatory syndrome, defined as an increase in CRP
  >10 mg/L).
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2016-02-06 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
NLR / CRP | 1 day
  To compare the NLR with other commonly used inflammatory markers for the diagnosis of bacterial infection in patients admitted for fever and/or inflammatory syndrome to an internal medicine department.
NLR / PCT | 1 day
  To compare the NLR with other commonly used inflammatory markers for the diagnosis of bacterial infection in patients admitted for fever and/or inflammatory syndrome to an internal medicine department.
NLR / white blood cell count | 1 day
  To compare the NLR with other commonly used inflammatory markers for the diagnosis of bacterial infection in patients admitted for fever and/or inflammatory syndrome to an internal medicine department.
NLR / PNN | 1 day
  To compare the NLR with other commonly used inflammatory markers for the diagnosis of bacterial infection in patients admitted for fever and/or inflammatory syndrome to an internal medicine department.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Schmidt, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens Picardie, Amiens, France